CLINICAL TRIAL: NCT07022470
Title: Brachytherapy Fractionation Individualized by Treatment Feasibility in Cervical Cancer: Phase II Trial Comparison of 3 vs 4 Fractions (BRACHY-FIT).
Brief Title: Phase II Trial Comparison of 3 vs 4 Fractions (BRACHY-FIT).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-79234
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancers
Keywords: high dose rate brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-Fraction Brachytherapy Arm (Experimental): Patients who meet dosimetric criteria at the first brachytherapy session (HR CTV D90 > 85 Gy and acceptable OAR constraints) will receive an investigational 3-fraction HDR brachytherapy regimen (24 Gy total).
  Interventions: Radiation: 3-Fraction HDR Brachytherapy
- Investigational Treatment (Active Comparator): Patients who do not meet dosimetric criteria for the investigational regimen will receive the institutional standard-of-care regimen of 4 fractions (28 Gy total).
  Interventions: Radiation: 4-Fraction HDR Brachytherapy

INTERVENTIONS:
Radiation: 3-Fraction HDR Brachytherapy — 8 Gy per fraction for 3 fractions (total 24 Gy) for patients with locally advanced cervical cancer, based on individualized planning.
  Arms: 3-Fraction Brachytherapy Arm
Radiation: 4-Fraction HDR Brachytherapy — 7 Gy per fraction for 4 fractions (total 28 Gy) as the standard-of-care brachytherapy regimen.
  Arms: Investigational Treatment

SUMMARY:
This is a prospective non-randomized clinical trial to evaluate the feasibility of 3 fraction versus a standard 4 fraction high dose rate brachytherapy regimen in patients with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented malignancy of the cervix and planned to receive brachytherapy as part of definitive treatment.
* ECOG performance status of 0-2
* Age ≥ 18 years old.
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Contraindication to receiving radiotherapy as determined by treating radiation oncologist.
* Contraindication to receiving MRI.
* Prior radiation to the pelvis > 3 months ago
* Age < 18 years old.
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Receiving 3-Fraction Brachytherapy Regimen | Up to 8 months
  Proportion of patients that underwent a 3 fraction brachytherapy regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States